CLINICAL TRIAL: NCT01971671
Title: Evaluation of the Nutrients Composition of Breast Milk of Chinese Lactating Mothers and Nutrition Intake of Chinese Pregnant and Lactating Mothers, Infants and Young Children
Brief Title: Evaluation of the Nutrients Composition of Breast Milk of Chinese Lactating Mothers and Their Nutrition Intake
Acronym: MING
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 11.14.NRC
Record Dates: First submitted 2013-10-14; First posted 2013-10-29 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Focus of Study is Healthy Chinese Lactating Mother 0-270 Days

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — breask milk sample.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chinese lactating mother: no intervention.
  Interventions: Other: no intervention.

INTERVENTIONS:
Other: no intervention.

SUMMARY:
To understand breast milk composition during different lactating stages.

ELIGIBILITY:
Inclusion Criteria:

* Chinese lactating mother 0-270 days after delivery (inclusive).
* Healthy with neither acute disease nor history of hereditary disease, gestational diabetes, hypertension, other concomitant diseases, and disability.
* Parents/ caregiver is willing to comply with the study procedure.
* Having received oral and written information about the aims and procedures of the study.
* Having obtained the her informed consent.

Exclusion Criteria:

* Subjects who are currently taking, or have taken in the last 4 weeks, or will take any medication.
* Subject who has history of psychopath and have no the dietary memory.
* Subjects who are suffering food allergy.
* Insufficient breast milk output according to the corresponding period after delivery.
* Alcoholic.
* Smokers.
* Subject who cannot be expected to comply with the study procedures.
* Currently participating or having participated in another clinical trial during the last 4 weeks prior to the beginning of this study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy Chinese lactating mother 0-270 days after delivery (inclusive) will be enrolled.
Sampling Method: Probability Sample
Enrollment: 560 (Actual)
Dates: Start 2011-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Primary outcome is the macronutrient composition of breast milk in Chinese lactating mothers from 0 to 270 days after delivery. | 0-270 days after delivery
  Macronutrient composition includes calories (kcal/ml), total protein, fat and carbohydrate (lactose) content in breast milk.

SECONDARY OUTCOMES:
Other nutrient composition in breast milk of 0-270 days after delivery. | 0-270 days after delivery.
  Beside macronutrient composition, all major minerals, vitamins will be analyzed. In addition, functional compounds, such as human milk oligosaccharides (HMOs), total/free amino acids, lipid profiles, and microbiota, will be analyzed as well.
Dietary pattern of lactating mothers of 0-270 days after delivery. | 0-270 days after delivery.
  A one-time standardized 24-hour food recall survey, is utilized to access dietary pattern of subjects.
Nutrients intake and adequacy of lactating mothers of 0-270 days after delivery. | 0-270 days after delivery
  A one-time standardized 24-hour food recall survey, is utilized to access nutrient intakes and adequacy (by comparing existing local and international RDAs and DRIs databases).
Nutrition supplements intake status of lactating mothers of 0-270 days after delivery. | 0-270 days after delivery.
  A one-time food frequency questionnaire (FFQ), designed to access nutritional supplement usage, is being utilized.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Science Center, Peking University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Xue Y, Redeuil KM, Gimenez EC, Vinyes-Pares G, Zhao A, He T, Yang X, Zheng Y, Zhang Y, Wang P, Thakkar SK. Regional, socioeconomic, and dietary factors influencing B-vitamins in human milk of urban Chinese lactating women at different lactation stages. BMC Nutr. 2017 Mar 7;3:22. doi: 10.1186/s40795-017-0139-1. eCollection 2017. PMID 32153804
- [Derived] Yu K, Xue Y, Zhao W, Zhao A, Li W, Zhang Y, Wang P. Translation of nutrient recommendations into personalized optimal diets for Chinese urban lactating women by linear programming models. BMC Pregnancy Childbirth. 2018 Sep 18;18(1):379. doi: 10.1186/s12884-018-2008-6. PMID 30227842